CLINICAL TRIAL: NCT05544448
Title: In Vitro Effect Study of Interleukin-2 Muteins on Regulatory T Cells of Patients With Different Autoimmune, Allo-immune or Inflammatory Diseases
Acronym: MuTreg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP220507
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases; Inflammatory Disease; Acquired Bone Marrow Aplasia; Systemic Lupus Erythematosus; Multiple Sclerosis; Gvhd; Rheumatoid Arthritis; Autoimmune Thyroiditis; Vitiligo; Alopecia; Atopic Dermatitis
Keywords: Autoimmune Diseases; Inflammation; Graft vs Host Disease; T-lymphocytes, Regulatory; Interleukin-2
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Multiple Sclerosis; Graft vs Host Disease; Arthritis, Rheumatoid; Thyroiditis, Autoimmune; Vitiligo; Alopecia; Dermatitis, Atopic; Inflammation

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, non-controlled, non-randomized in vitro study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample taken at a single time point — At inclusion, a blood sample will be taken for research purpose

SUMMARY:
Interleukin 2 (IL-2) is a critical cytokine for the survival and function of regulatory T cells (LTreg). This cytokine has a dual role in the immune system. IL-2 stimulates immune responses by acting on the intermediate affinity IL-2R receptor, IL-2Rβγ, expressed by conventional T cells (LTconv) during activation, but also contributes to the inhibition of immune responses via LTreg that express the high affinity receptor IL-2Rαβγ.

This difference in IL-2 receptor affinity for IL-2 has led to the development of low-dose IL-2 therapy to stimulate LTreg and improve control of excessive inflammation in autoimmune (AID), inflammatory or alloimmune diseases Low-dose IL-2 therapy is being studied in several of these diseases such as systemic lupus erythematosus, type 1 diabetes, alopecia, HCV (hepatitis C virus)-induced vasculitis, atopic dermatitis and chronic allo-transplantation-related graft-versus-host disease (GVHD).

Some of these studies have shown an increase in LTreg numbers and an improvement in certain clinical signs.

To improve LTreg targeting in autoimmune diseases, inflammatory diseases or GVHD, mutated IL-2s (muteins) have been developed with selective LTreg agonist properties.

These IL-2 muteins are linked to an Fc fragment to increase their half-life. Two IL-2 variants (IL-2Vs)-Fc preferentially stimulate STAT5 phosphorylation in LTregs compared to conventional FoxP3- (LTconv) CD4+ or CD8+ T cells

DETAILED DESCRIPTION:
Hypothesis:

In order to confirm that this differential effect of IL-2 muteins, already established in non-diseased controls, is also observed in patients with autoimmune diseases, inflammatory diseases or GVHD, a pilot in vitro study should be conducted on a small number of patient's blood samples (5 or 10 depending on the pathology).

Objective :

Conduct a multicentre pilot study to confirm the hypothesis that IL-2 muteins preferentially activate the STAT5 pathway in LTreg compared to LTconv in patients with GVHD, acquired bone marrow aplasia, systemic lupus erythematosus, multiple sclerosis, rheumatoid arthritis, autoimmune thyroiditis, vitiligo, alopecia or atopic dermatitis

Method:

At the inclusion, patients will have a blood sample collected for in vitro research purposes. Their clinical data will also be collected.

Conclusion This trial should provide in vitro proof-of-principle of the efficacy of IL-2 muteins on LTreg and could eventually lead to a therapeutic trial

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria common to all patients in different departments:
* Age18 years
* Affiliated to social security or entitled to
* Patient who has been informed of the study and has signed a free and informed consent

Inclusion criteria specific by department:

Inclusion criteria for Clinical Hematology Department:

* Patient with GVHD following allogeneic hematopoietic stem cell transplantation (HSC)
* Or with acquired bone marrow suppression
* Lymphocytosis > 0.5 G/L

Inclusion criteria for Nephrology and Transplantation department:

- Patient with systemic lupus erythematosus (ACR classification criteria)

Inclusion criteria for Neurology department:

- Patient with multiple sclerosis (criteria of Mc Donald 2017)

Inclusion criteria for Rheumatology Department:

- Patient with rheumatoid arthritis (ACR classification criteria)

Inclusion criteria for Internal Medicine-Endocrinology Department:

- Patient with Basedow disease, Hashimoto's thyroiditis

Inclusion criteria for Dermatology Department:

- Patient with vitiligo or alopecia areata or atopic dermatitis

Exclusion Criteria:

Non-inclusion criteria common to all patients:

* Patient under guardianship, curatorship or judicial protection
* Pregnant, parturient or breastfeeding woman
* Patient deprived of liberty
* Patient hospitalized without consent
* Patient admitted to a health or social institution for purposes other than research
* Minor patient
* Adult patient unable to express consent
* Refusal to participate
* Patient on AME

Non-inclusion criteria specific by department:

Non-inclusion criteria for Clinical Hematology Department:

* Ongoing treatment with high doses (>1 mg/kg/d) of systemic corticosteroid therapy
* Ongoing treatment with JAK inhibitors

Non-inclusion criteria for Nephrology and Transplantation Department:

* Ongoing treatment with doses >10 mg/d Prednisone
* Ongoing treatment with Cellcept, Endoxan, Imurel, Belimumab, Anti-CD20, Methotrexate
* Ongoing treatment with JAK inhibitors

Non-inclusion criteria for Neurology Department:

* Treatment with systemic corticosteroid therapy, Fingolimod or Teriflunomide
* Ongoing treatment with JAK inhibitors
* Lymphocytosis < 0.5 G/L

Non-inclusion criteria for Rheumatology Department:

* Ongoing treatment with doses >15 mg/d Prednisone
* Treatment with Rituximab or Tocilizumab
* Ongoing treatment with JAK inhibitors
* Lymphocytosis < 0.5 G/L

Non-inclusion criteria for Internal Medicine - Endocrinology Department:

* Ongoing immunosuppressive therapy
* Ongoing treatment with JAK inhibitors

Non-inclusion criteria for Dermatology Department:

* Ongoing treatment with Methotrexate
* Ongoing treatment with JAK inhibitors
* Ongoing treatment with doses >10 mg/d prednisone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
the percentage of phosphorylated STAT5 in LTresg compared to LTconv after incubation with IL-2 muteins | At inclusion
  The measurement method is based on the quantification of the phosphorylated STAT5 molecule in LTconv and LTreg by flow cytometry after incubating the cells with IL-2 or IL-2 muteins

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, 1 rue Gustave Eiffel,, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No